CLINICAL TRIAL: NCT06750757
Title: Intraoperative Bone Marrow Aspirate Concentrate Injections: Evaluating Outcomes in a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: American Hip Institute (Other)
Responsible Party: Principal Investigator, Benjamin Domb, MD, Medical Director, American Hip Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHI-006
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Labral Tear; Femoroacetabular Impingement
Keywords: hip arthroscopy; bone marrow aspirate concentrate; orthobiologics
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BMAC Arm (Experimental)
  Interventions: Biological: Bone marrow aspirate concentrate; Procedure: Hip arthroscopy
- No BMAC (Control) (Active Comparator)
  Interventions: Procedure: Hip arthroscopy

INTERVENTIONS:
Biological: Bone marrow aspirate concentrate — 145cc of BMAC/PRP/PPP injection.
  Other Names: BMAC
  Arms: BMAC Arm
Procedure: Hip arthroscopy — Both groups will undergo a hip arthroscopy to treat their condition. However, the control group will not receive a BMAC injection during the surgery.

SUMMARY:
The purpose of this study is to see if bone marrow aspirate concentrate (BMAC) used with your hip arthroscopy surgery is a better treatment than just having surgery alone for treatment of labral tears in your hip.

BMAC is an injection, where your doctor will insert a needle into your hip and harvest the bone marrow that is located inside of your bones. This will be performed under anesthesia during your hip arthroscopy surgery and will be injected during the procedure. BMAC is an FDA approved procedure and has had many research articles produced from it.

Researchers will compare patients who received BMAC during their surgery to those who have not to determine if the injection with surgery is better than surgery alone.

DETAILED DESCRIPTION:
Background and Significance Hip pain and dysfunction are common ailments in the adult population that deleteriously impact sport participation, recreational hobbies, activities of daily living, and often the ability to earn a living. Femoroacetabular impingement (FAI) with labral tearing is a leading cause of pre-arthritic hip pain that is often treated with hip arthroscopy and labral repair. There have been significant advances in techniques utilized to treat the labrum, including segmental and circumferential reconstruction, as well as the hip capsule, including repair, plication, and reconstruction. These modern techniques have resulted in durable therapeutic gain with largely successful outcomes 10 years postoperatively. Despite these advances, severe cartilage injury diagnosed intraoperatively is associated with inferior outcomes and higher rates of short- and long-term conversion to total hip arthroplasty. Further, treatment options for acetabular and femoral head chondral damage are limited, with microfracture serving as the current standard of care.

Innovations in regenerative medicine including platelet-rich-plasma (PRP), as well as cell-based therapies including bone marrow aspirate concentrate (BMAC) have received increasing attention in both the academic and general populations. While isolated intraoperative PRP application has not shown significant benefit, multiple studies have shown promising outcomes following intraoperative e application of BMAC during hip arthroscopy for FAI. A 2021 report by Martin and colleagues found significantly improved two-year postoperative outcomes in patients with Outerbridge grade II/III acetabular chondral defects that received intraoperative BMAC compared to a matched historical control group. These findings have been reinforced by subsequent studies demonstrating superiority of BMAC compared to microfracture as well as similar patient reported outcomes in patients with Tonnis radiographic grade I-II osteoarthritis who received BMAC when compared to a non-arthritic cohort. Taken together, these recent findings suggest that intraoperative BMAC application can improve outcomes following hip arthroscopy for FAI, particularly in the setting of cartilage damage and early arthritis. To date, no level one study has evaluated the impact of intraoperative BMAC on patient outcomes following hip arthroscopy for FAI. Given the absence of available high quality literature, a blinded, randomized controlled trial Given the cost, as well as potential bias associated with BMAC application a blinded

Design & Methods Study Design The proposed study has received institutional review board approval and is currently in the registration process for randomized controlled trials at clinicaltrials.gov. The study will consist of subjects undergoing hip arthroscopy for femoroacetabular impingement that will be randomized to receive a single intraoperative BMAC/PRP injection. BMAC will be harvested through the standard arthroscopic portals adopting the methodology reported by Martin et al. allowing for patient blinding to treatment. The surgeon will not be blinded to treatment administered at the time of the procedure, however data analysis will be performed by institutional staff blinded to subject treatment arms. The study goals and methodology will be discussed with potential candidates and informed consent will be obtained in the office during the preoperative appointment. Covariate adaptive randomization will occur prior to surgery with the goal of minimizing preoperative demographic and radiographic differences between the BMAC and control group. An a priori power analysis was constructed using the international hip outcome tool (iHOT-12) minimum clinically important difference (MCID) of 13 points, a score standard deviation of 18, and an α error of 0.05, which determined 32 subjects in each group would be required to achieve sufficient power (1-β) of 80%. To allow for a 20% drop out rate, the study goal is to obtain a minimum of 40 patients for each group.

Study Methodology Study inclusion criteria will consist of patients undergoing primary hip arthroscopy to treat femoroacetabular impingement. Subjects will require a clinical diagnosis of intra-articular pathology consisting of anterior hip and/or groin pain with restricted hip motion and positive impingement testing. Study inclusion also requires the radiographic hallmarks of Cam type femoroacetabular impingement with an alpha angle greater than 60 degrees on Dunn lateral views and advanced imaging with magnetic resonance imaging (MRI) or magnetic resonance arthrography (MRA) confirming chondrolabral pathology. Subjects will be excluded if they have had prior hip arthroscopy or hip surgery, Tonnis grade II or higher radiographic osteoarthritis, congenital hip deformities including Legg-Calve-Perthes or Slipped Capital Femoral Epiphysis, rheumatologic conditions, or workers compensation claims. Patients undergoing additional arthroscopic procedures such as trochanteric bursectomy or gluteus medius repair will also be excluded.

Potential subjects will then be introduced to the study by the treating surgeon, and if interested will discuss the study further with institutional staff. Subjects will be educated on the intraoperative harvest and application of BMAC as well as potential risks and benefits of the procedure. Given that the patient is under general anesthesia for the hip arthroscopy procedure, and no additional portals or incisions are created, additional risks related to harvest are considered minimal. Patients interested in participating in the study will be instructed that they will be randomized prior to their surgery and that they may or may not receive BMAC treatment depending on the results of the randomization. Patients that are not interested in participating in the study will still be offered intraoperative BMAC application but will be instructed that this will occur as an out-of-pocket expense. The patient will then be formally consented for the study by office staff. Randomization will be carried out according to the covariate adaptive methodology described by Frane et al to minimize potential demographic and radiographic differences between groups, with the designated treatment group sealed in an envelope to be opened at the time of surgery.

Preoperative data acquisition:

Preoperative patient data collection will include age, gender, body mass index (BMI), and Beighton's score, with radiographic variables including the alpha angle, lateral center edge angle (LCEA), anterior center edge angle (ACEA), alpha angle, Tonnis grade, and joint space width. Advanced imaging with 3-D computed tomography (CT) reconstruction will include measurements of acetabular and femoral version while magnetic resonance imaging will be graded according the Scoriing of Hip Osteoarthritis in MRI (SHOMRI) classification. The SHOMRI classification is a validated semi-quantitative grading system to evaluate chondrolabral damage as well as other markers of osteoarthritis on MRI including subchondral cystic change, subchondral edema, loose bodies, and joint effusions. The SHOMRI classification has subsequently shown significant correlations to arthroscopic findings as well as demonstrated the ability to detect change with disease progression (Schwaiger, Heerey).

Surgical Procedure Hip arthroscopy for FAI will be performed on all patients included in the study. Briefly, following induction of general anesthesia, patients will be placed supine on an operative table designed for hip arthroscopy. Before positioning, 51cc of whole blood will be drawn with 8cc of normal saline and 1cc of anticoagulant citrate dextrose solution A (ACD-A), and centrifuged according to the manufacturer's instructions (Angel PRP, Arthrex, Naples, FL) to obtain a combination of platelet rich plasma (PRP) and platelet poor plasma (PPP). The PRP and PPP will then be combined to form a PPP/PRP mixture and placed in a sterile cup on the operating table. Hip joint access will be established under fluoroscopic guidance following the application of traction. A diagnostic arthroscopy will be performed to determine the extent of intra-articular pathology. Specific intraoperative findings that are recorded include the labrum tear type (Seldes) and length, and femoral head and acetabular chondral pathology will be diagnosed according to the Outerbridge grading scale. Ligamentum Teres damage will be classified according to the Domb and Villar grading scales.

Following diagnostic arthroscopy, BMAC harvest will be performed according to the technique described by Martin et al. Viewing through the mid-anterior portal, a 15-guage Jamshidi bone marrow biopsy aspiration needle will be placed to access the ilium under a combination of fluoroscopic guidance and arthroscopic visualization. The access point is proximal to the sourcil and lateral to the reflected head of the rectus. Once the access point has been identified, the needle is malleted through the outer cortex of the ilium and guided 1cm medially under fluoroscopic guidance. According to the manufacturer's protocol, a heparin rinsed syringe is attached and bone marrow is aspirated under gentle negative pressure with the goal of harvesting 75cc of blood product for downstream processing. Following harvest, the bone marrow aspirate is then centrifuged to obtain BMAC which is then aseptically transferred to the previously obtained PRP/PPP mixture. During processing, the remainder of the indicated procedures are carried out including labral treatment with repair or reconstruction, chondroplasty, ligamentum teres debridement, acetabuloplasty, and femoroplasty. In cases of full thickness (Outerbridge grade IV) cartilage damage, the lesion will be treated with debridement and abrasion without microfracture. Following completion of the femoroplasty, the BMAC/PRP/PPP slurry will then be combined with 10,000U thrombin in 10cc of saline to begin the clotting cascade several minutes prior to application. The product will then be transferred to a syringe and injected into the central compartment under direct arthroscopic visualization with the inflow switched off. The hip is then reduced and flexed to 45 degrees with confirmation of the product remaining in the central compartment prior to the re-establishment of fluid flow. The hip capsule is then closed using absorbable interrupted vicryl sutures and the portals closed with interrupted nylon sutures.

Rehabilitation A previously reported 4-phase rehabilitation program will begin on post-operative day one for all patients. Briefly, patients will be foot flat weight-bearing in a postoperative hip brace for two weeks for labral repairs and six weeks for labral reconstructions. There is no difference in rehabilitation protocol between the treatment groups.

Outcome assessment Patients will receive follow-up at the 2-week, 6-week, 4 month, 7 month, and one year time point followed by annual follow-up thereafter completed either in the office or electronically for evaluation of patient reported outcome measures (PROMs). Clinical outcome analysis will include complications as well as reoperation for revision arthroscopy, revision open hip preservation surgery, or hip reconstruction surgery. Patient reported outcomes will include the iHOT-12 as the primary outcome measure with the modified Harris Hip Score (mHHS), non-arthritic hip score (NAHS), Hip Outcome Score-Sports Subscale (HOS-SSS) and Visual Analog Scale for pain (VAS) as secondary outcome measures. The MCID and the patient acceptable symptomatic state (PASS) for each PROMS will be the two primary clinically relevant outcome thresholds evaluated in this study.

Statistical Analysis Continuous variables will be tested for normality and variance using the Shapiro-Wilk test and F test respectively. Continuous variables will then be compared between groups using parametric t-tests or one-way analysis of variance (ANOVA), or non-parametric Mann-Whitney U or Welch tests where appropriate. Categorical variables will be compared using the Pearson chi-square or Fischer exact test. The MCID will be calculated for each group according to the ½ standard deviation approach described by Normal et al, while the PASS threshold will be calculated for each group using the Youden index to optimize the sensitivity and specificity parameters for each outcome survey with respect to the anchor-based PASS methodology. Nominal logistic multivariate regression will then be performed to identify factors predictive of achieving clinically relevant outcome thresholds. A p-value of 0.05 will be used to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary hip arthroscopy to treat femoroacetabular impingement
* Subjects will require a clinical diagnosis of intra-articular pathology consisting of anterior hip and/or groin pain with restricted hip motion and positive impingement testing.
* Study inclusion also requires the radiographic hallmarks of Cam type femoroacetabular impingement with an alpha angle greater than 60 degrees on Dunn lateral views and advanced imaging with magnetic resonance imaging (MRI) or magnetic resonance arthrography (MRA) confirming chondrolabral pathology.

Exclusion Criteria:

* Patients who have had prior hip arthroscopy or hip surgery, Tonnis grade II or higher radiographic osteoarthritis, congenital hip deformities including Legg-Calve-Perthes or Slipped Capital Femoral Epiphysis, rheumatologic conditions, or workers compensation claims.
* Patients undergoing additional arthroscopic procedures such as trochanteric bursectomy or gluteus medius repair will also be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
iHOT-12 | 2 years

SECONDARY OUTCOMES:
modified Harris Hip Score | 2 years
Non-arthritic hip score | 2 years
Hip outcome score-sports specific subscale | 2 years
Visual analog scale | 2 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan JJ, Vogel MJ, Larson JH, Nho SJ. Cartilage Defects Are Negatively Associated With Long-Term Hip Survivorship Following Contemporary Hip Arthroscopy for Femoroacetabular Impingement Syndrome: A Propensity-Matched Analysis at Minimum 10-Year Follow-Up. Arthroscopy. 2024 Nov;40(11):2681-2692. doi: 10.1016/j.arthro.2024.01.040. Epub 2024 Feb 7. PMID 38331365
- [Background] MacDonald AE, Bedi A, Horner NS, de Sa D, Simunovic N, Philippon MJ, Ayeni OR. Indications and Outcomes for Microfracture as an Adjunct to Hip Arthroscopy for Treatment of Chondral Defects in Patients With Femoroacetabular Impingement: A Systematic Review. Arthroscopy. 2016 Jan;32(1):190-200.e2. doi: 10.1016/j.arthro.2015.06.041. Epub 2015 Sep 15. PMID 26385287
- [Background] George T, Curley AJ, Saeed SK, Kuhns BD, Parsa A, Domb BG. Orthobiologics as an adjunct in treatment of femoroacetabular impingement syndrome: cell-based therapies facilitate improved postoperative outcomes in the setting of acetabular chondral lesions-a systematic review. Knee Surg Sports Traumatol Arthrosc. 2023 Dec;31(12):6020-6038. doi: 10.1007/s00167-023-07624-4. Epub 2023 Oct 31. PMID 37906291
- [Background] Siddiq BS, Giorgino R, Gillinov SM, Lee JS, Dowley KS, Cherian NJ, Martin SD. Neither Bone Marrow Aspirate Concentrate nor Platelet-Rich Plasma Improves Patient-Reported Outcomes After Surgical Management of Acetabular Labral Tears; However, Bone Marrow Aspirate Concentrate May Be Effective for Moderate Cartilage Damage: A Systematic Review. Arthrosc Sports Med Rehabil. 2024 Aug 28;6(6):100991. doi: 10.1016/j.asmr.2024.100991. eCollection 2024 Dec. PMID 39776509
- [Background] Kucharik MP, Abraham PF, Nazal MR, Varady NH, Eberlin CT, Meek WM, Naessig SA, Martin SD. Treatment of Full-Thickness Acetabular Chondral Flaps During Hip Arthroscopy: Bone Marrow Aspirate Concentrate Versus Microfracture. Orthop J Sports Med. 2021 Dec 7;9(12):23259671211059170. doi: 10.1177/23259671211059170. eCollection 2021 Dec. PMID 34901293
- [Background] Bodendorfer BM, DeFroda SF, Clapp IM, Newhouse A, Nwachukwu BU, Nho SJ. Defining Clinically Significant Improvement on the Patient-Reported Outcomes Measurement Information System Test at 1-Year Follow-up for Patients Undergoing Hip Arthroscopy for the Treatment of Femoroacetabular Impingement Syndrome. Am J Sports Med. 2021 Jul;49(9):2457-2465. doi: 10.1177/03635465211015687. Epub 2021 Jun 7. PMID 34097552
- [Background] Frane JW. A Method of Biased Coin Randomization, Its Implementation, and Its Validation. Drug Inf J : DIJ Drug Inf Assoc 1998;32:423-32. https://doi.org/10.1177/009286159803200213.
- [Background] Li X, Zhou J, Hu F. Testing hypotheses under adaptive randomization with continuous covariates in clinical trials. Stat Methods Med Res. 2019 Jun;28(6):1609-1621. doi: 10.1177/0962280218770231. Epub 2018 May 17. PMID 29770730
- [Background] Lee S, Nardo L, Kumar D, Wyatt CR, Souza RB, Lynch J, McCulloch CE, Majumdar S, Lane NE, Link TM. Scoring hip osteoarthritis with MRI (SHOMRI): A whole joint osteoarthritis evaluation system. J Magn Reson Imaging. 2015 Jun;41(6):1549-57. doi: 10.1002/jmri.24722. Epub 2014 Aug 20. PMID 25139720
- [Background] Grace T, Neumann J, Samaan MA, Souza RB, Majumdar S, Link TM, Zhang AL. Using the Scoring Hip Osteoarthritis with Magnetic Resonance Imaging (SHOMRI) system to assess intra-articular pathology in femoroacetabular impingement. J Orthop Res. 2018 Nov;36(11):3064-3070. doi: 10.1002/jor.24102. Epub 2018 Jul 13. PMID 29947434
- [Background] Neumann J, Zhang AL, Schwaiger BJ, Samaan MA, Souza R, Foreman SC, Joseph GB, Grace T, Majumdar S, Link TM. Validation of scoring hip osteoarthritis with MRI (SHOMRI) scores using hip arthroscopy as a standard of reference. Eur Radiol. 2019 Feb;29(2):578-587. doi: 10.1007/s00330-018-5623-8. Epub 2018 Jul 9. PMID 29987419
- [Background] Heerey JJ, Souza RB, Link TM, Luitjens J, Gassert F, Kemp JL, Scholes MJ, Crossley KM. Defining hip osteoarthritis feature prevalence, severity, and change using the Scoring of Hip Osteoarthritis with MRI (SHOMRI). Skeletal Radiol. 2024 Aug;53(8):1599-1609. doi: 10.1007/s00256-024-04628-0. Epub 2024 Mar 9. PMID 38459982
- [Background] Schwaiger BJ, Gersing AS, Lee S, Nardo L, Samaan MA, Souza RB, Link TM, Majumdar S. Longitudinal assessment of MRI in hip osteoarthritis using SHOMRI and correlation with clinical progression. Semin Arthritis Rheum. 2016 Jun;45(6):648-55. doi: 10.1016/j.semarthrit.2016.04.001. Epub 2016 Apr 8. PMID 27162009
- [Background] Maldonado DR, Rosinsky PJ, Shapira J, Domb BG. Stepwise Safe Access in Hip Arthroscopy in the Supine Position: Tips and Pearls From A to Z. J Am Acad Orthop Surg. 2020 Aug 15;28(16):651-659. doi: 10.5435/JAAOS-D-19-00856. PMID 32769716
- [Background] Seldes RM, Tan V, Hunt J, Katz M, Winiarsky R, Fitzgerald RH Jr. Anatomy, histologic features, and vascularity of the adult acetabular labrum. Clin Orthop Relat Res. 2001 Jan;(382):232-40. doi: 10.1097/00003086-200101000-00031. PMID 11153993
- [Background] Outerbridge RE. The etiology of chondromalacia patellae. 1961. Clin Orthop Relat Res. 2001 Aug;(389):5-8. doi: 10.1097/00003086-200108000-00002. No abstract available. PMID 11501822
- [Background] Botser IB, Martin DE, Stout CE, Domb BG. Tears of the ligamentum teres: prevalence in hip arthroscopy using 2 classification systems. Am J Sports Med. 2011 Jul;39 Suppl:117S-25S. doi: 10.1177/0363546511413865. PMID 21709041
- [Background] Domb BG, Sgroi TA, VanDevender JC. Physical Therapy Protocol After Hip Arthroscopy: Clinical Guidelines Supported by 2-Year Outcomes. Sports Health. 2016 Jul;8(4):347-54. doi: 10.1177/1941738116647920. Epub 2016 May 12. PMID 27173983
- [Background] Chahal J, Van Thiel GS, Mather RC 3rd, Lee S, Song SH, Davis AM, Salata M, Nho SJ. The Patient Acceptable Symptomatic State for the Modified Harris Hip Score and Hip Outcome Score Among Patients Undergoing Surgical Treatment for Femoroacetabular Impingement. Am J Sports Med. 2015 Aug;43(8):1844-9. doi: 10.1177/0363546515587739. Epub 2015 Jun 15. PMID 26078452
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state. Ann Rheum Dis. 2005 Jan;64(1):34-7. doi: 10.1136/ard.2004.023028. Epub 2004 May 6. PMID 15130902
- [Background] Zusmanovich M, Haselman W, Serrano B, Banffy M. The Incidence of Hip Arthroscopy in Patients With Femoroacetabular Impingement Syndrome and Labral Pathology Increased by 85% Between 2011 and 2018 in the United States. Arthroscopy. 2022 Jan;38(1):82-87. doi: 10.1016/j.arthro.2021.04.049. Epub 2021 May 5. PMID 33964383
- [Background] Griffin DR, Dickenson EJ, O'Donnell J, Agricola R, Awan T, Beck M, Clohisy JC, Dijkstra HP, Falvey E, Gimpel M, Hinman RS, Holmich P, Kassarjian A, Martin HD, Martin R, Mather RC, Philippon MJ, Reiman MP, Takla A, Thorborg K, Walker S, Weir A, Bennell KL. The Warwick Agreement on femoroacetabular impingement syndrome (FAI syndrome): an international consensus statement. Br J Sports Med. 2016 Oct;50(19):1169-76. doi: 10.1136/bjsports-2016-096743. PMID 27629403
- [Background] Ibarra C, Villalobos E, Madrazo-Ibarra A, Velasquillo C, Martinez-Lopez V, Izaguirre A, Olivos-Meza A, Cortes-Gonzalez S, Perez-Jimenez FJ, Vargas-Ramirez A, Franco-Sanchez G, Ibarra-Ibarra LG, Sierra-Suarez L, Almazan A, Ortega-Sanchez C, Trueba C, Martin FB, Arredondo-Valdes R, Chavez-Arias D. Arthroscopic Matrix-Assisted Autologous Chondrocyte Transplantation Versus Microfracture: A 6-Year Follow-up of a Prospective Randomized Trial. Am J Sports Med. 2021 Jul;49(8):2165-2176. doi: 10.1177/03635465211010487. Epub 2021 May 28. PMID 34048286
- [Background] Bretschneider H, Trattnig S, Landgraeber S, Hartmann A, Gunther KP, Dienst M, Schroder J, Fickert S. Arthroscopic matrix-associated, injectable autologous chondrocyte transplantation of the hip: significant improvement in patient-related outcome and good transplant quality in MRI assessment. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1317-1324. doi: 10.1007/s00167-019-05466-7. Epub 2019 Apr 16. PMID 30993353
- [Background] Gebhardt S, Hofer A, Wassilew GI, Sobau C, Zimmerer A. Minced Cartilage Implantation in Acetabular Cartilage Defects: Case Series with 2-Year Results. Cartilage. 2023 Dec;14(4):393-399. doi: 10.1177/19476035231189840. Epub 2023 Aug 3. PMID 37533396
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681
- [Background] Stelzer JW, Martin SD. Use of Bone Marrow Aspirate Concentrate with Acetabular Labral Repair for the Management of Chondrolabral Junction Breakdown. Arthrosc Tech. 2018 Sep 1;7(10):e981-e987. doi: 10.1016/j.eats.2018.06.003. eCollection 2018 Oct. PMID 30377577
- [Background] Martin SD, Eberlin CT, Kucharik MP, Cherian NJ. Harvest and Application of Bone Marrow Aspirate Concentrate to Address Acetabular Chondral Damage During Hip Arthroscopy. JBJS Essent Surg Tech. 2023 May 24;13(2):e22.00010. doi: 10.2106/JBJS.ST.22.00010. eCollection 2023 Apr-Jun. PMID 38274149
- [Background] Sullivan SW, Aladesuru OM, Ranawat AS, Nwachukwu BU. The use of biologics to improve patient-reported outcomes in hip preservation. J Hip Preserv Surg. 2021 Apr 17;8(1):3-13. doi: 10.1093/jhps/hnab028. eCollection 2021 Jan. PMID 34567595
- [Background] Hevesi M, Jacob G, Shimomura K, Ando W, Nakamura N, Krych AJ. Current hip cartilage regeneration/repair modalities: a scoping review of biologics and surgery. Int Orthop. 2021 Feb;45(2):319-333. doi: 10.1007/s00264-020-04789-2. Epub 2020 Sep 10. PMID 32910240
- [Background] Jildeh TR, Abbas MJ, Buckley P, Okoroha KR. The Use of Biologics for Hip Preservation. Curr Rev Musculoskelet Med. 2021 Apr;14(2):145-154. doi: 10.1007/s12178-021-09695-7. Epub 2021 Jan 23. PMID 33483876
- [Background] Kim DN, Fong S, Park N, Simington J, Atadja L, Pettinelli N, Lee MS, Gillinov SM, Maldonado DR, Jimenez AE. Mid- to Long-Term Outcomes in Patients After Hip Arthroscopy With Labral Reconstruction: A Systematic Review. Orthop J Sports Med. 2024 Jun 1;12(6):23259671241232306. doi: 10.1177/23259671241232306. eCollection 2024 Jun. PMID 38831872
- [Background] Philippon MJ, Arner JW, Crawford MD, Bolia IK, Briggs KK. Acetabular Labral Reconstruction with Iliotibial Band Autograft: Outcome and Survivorship at a Minimum 10-Year Follow-up. J Bone Joint Surg Am. 2020 Sep 16;102(18):1581-1587. doi: 10.2106/JBJS.19.01499. PMID 32675477
- [Background] Ganz R, Parvizi J, Beck M, Leunig M, Notzli H, Siebenrock KA. Femoroacetabular impingement: a cause for osteoarthritis of the hip. Clin Orthop Relat Res. 2003 Dec;(417):112-20. doi: 10.1097/01.blo.0000096804.78689.c2. PMID 14646708
- [Background] Rivera E, Seijas R, Rubio M, Garcia-Balletbo M, Vilar JM, Boada PL, Cugat R. Outcomes at 2-Years Follow-Up After Hip Arthroscopy Combining Bone Marrow Concentrate. J Invest Surg. 2020 Aug;33(7):655-663. doi: 10.1080/08941939.2018.1535010. Epub 2019 Apr 7. PMID 30957569
- [Background] Day MA, Hancock KJ, Selley RS, Olsen R, Ranawat AS, Nwachukwu BU, Kelly BT, Nawabi DH. Hip Arthroscopy With Bone Marrow Aspirate Injection for Patients With Symptomatic Labral Tears and Early Degenerative Changes Shows Similar Improvement Compared With Patients Undergoing Hip Arthroscopy With Symptomatic Labral Tears Without Arthritis. Arthroscopy. 2023 Jun;39(6):1429-1437. doi: 10.1016/j.arthro.2022.12.012. Epub 2022 Dec 24. PMID 36574821
- [Background] Martin SD, Kucharik MP, Abraham PF, Nazal MR, Meek WM, Varady NH. Functional Outcomes of Arthroscopic Acetabular Labral Repair with and without Bone Marrow Aspirate Concentrate. J Bone Joint Surg Am. 2022 Jan 5;104(1):4-14. doi: 10.2106/JBJS.20.01740. PMID 34648479
- [Background] Menge TJ, Briggs KK, Dornan GJ, McNamara SC, Philippon MJ. Survivorship and Outcomes 10 Years Following Hip Arthroscopy for Femoroacetabular Impingement: Labral Debridement Compared with Labral Repair. J Bone Joint Surg Am. 2017 Jun 21;99(12):997-1004. doi: 10.2106/JBJS.16.01060. PMID 28632588
- [Background] Dwyer MK, Tumpowsky C, Boone A, Lee J, McCarthy JC. What Is the Association Between Articular Cartilage Damage and Subsequent THA 20 Years After Hip Arthroscopy for Labral Tears? Clin Orthop Relat Res. 2019 May;477(5):1211-1220. doi: 10.1097/CORR.0000000000000717. PMID 30998639
- [Background] Dwyer MK, Lee JA, McCarthy JC. Cartilage Status at Time of Arthroscopy Predicts Failure in Patients With Hip Dysplasia. J Arthroplasty. 2015 Sep;30(9 Suppl):121-4. doi: 10.1016/j.arth.2014.12.034. Epub 2015 Jun 3. PMID 26059500
- [Background] Suarez-Ahedo C, Gui C, Rabe SM, Chandrasekaran S, Lodhia P, Domb BG. Acetabular Chondral Lesions in Hip Arthroscopy: Relationships Between Grade, Topography, and Demographics. Am J Sports Med. 2017 Sep;45(11):2501-2506. doi: 10.1177/0363546517708192. Epub 2017 Jun 7. PMID 28590784